CLINICAL TRIAL: NCT01055379
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate if Rasagiline Can Improve Depressive Symptoms and Cognitive Function in Non-demented, Idiopathic Parkinson's Disease Patients: ACCORDO Study
Brief Title: Rasagiline in Cognitive-impairment Related Depression: AzileCt in COgnitive-impairment Related DepressiOn
Acronym: ACCORDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundbeck Italia S.p.A. (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12962A; 2009-011144-19 (EudraCT Number)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Depressive Symptoms; Parkinson's Disease
Keywords: Rasagiline; Depressive Symptoms; Cognition
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline (Experimental)
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — 1 mg/day for 12 weeks; orally
  Other Names: Azilect
  Arms: Rasagiline
Drug: Placebo — Once daily for 12 weeks; orally
  Arms: Placebo

SUMMARY:
The primary endpoint for this study is the clinical response after 12 weeks of treatment, defined as a change in total score from baseline depressive symptoms as measured by the Beck Depression Inventory-Amended (BDI-IA) total score.

DETAILED DESCRIPTION:
ACCORDO is a multicentre, randomised, double-blind, and placebo-controlled study conducted in 12 Italian centres. Subjects are screened by means of the BDI-IA (cut-off 15) and randomised to treatment with rasagiline or placebo for 12 weeks.

Subjects have to be on stable treatment with dopaminergic agents at least 4 weeks before baseline, and maintained so during the course of the study.

The primary objective is to evaluate whether rasagiline compared to placebo improves depressive symptoms as evaluated by the BDI-IA total score.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female aged >=40 and <80 years. The subject has a diagnosis of idiopathic Parkinson's Disease (PD) according to the United Kingdom Parkinson's Disease Society brain bank diagnostic criteria for PD for the clinical diagnosis of PD.
* Depressive symptoms with a minimum severity of >=15 using the BDI-IA.
* Hoehn and Yahr stage I-III.
* Under stable (4 weeks prior to baseline) dopaminergic treatment without significant motor complication such as "on-off" phenomena and/or dyskinesia.
* The subject and/or legal representative and/or impartial witness is/are able to read and understand the Subject Information Sheet.
* The subject and/or legal representative has/have signed the Informed Consent Form (ICF) and if relevant the impartial witness has co-signed the ICF.
* If female, must: agree not to try to become pregnant during the study (female patients of childbearing potential will take pregnancy test, using a urine stick), AND use adequate contraception (adequate contraception is defined as oral/systemic contraception, intrauterine device, diaphragm in combination with spermicidal, or condom for male partner in combination with spermicidal), OR have been menopausal for at least 24 months prior to baseline, (OR) have been surgically sterilised prior to baseline, OR have had a hysterectomy prior to baseline.

Exclusion Criteria:

A subject, who meets one or more of the following criteria at the Baseline Visit, is not eligible for inclusion in this study:

* Motor complications such as wearing off and on-off phenomena.
* Mini-Mental State Examination (MMSE) <26, corrected score.
* Diagnosis of current or history of major depressive episode according to DSM-IV-TR® criteria within 1 year before recruitment into the study.
* Presence of any other neurodegenerative disorder other than PD, based on judgement of investigator.
* Psychotic symptoms, e.g. hallucination and delirium (determined by clinical evaluation).
* Presence of any unstable or untreated systemic disorder such as diabetes, cardiac failure, or renal failure.
* Use of any prohibited concomitant medication according to the timelines provided in Appendix II.
* Patient who have undergone Deep Brain Stimulation surgery.
* Current treatment with antidepressants or history of treatment with antidepressants less than 1 month prior to randomisation.
* Current treatment or history of treatment less than 1 month prior to randomisation, with antipsychotics, cholinesterase inhibitors, memantine, amantadine, or anticholinergics.
* Current treatment with selegiline or history of treatment with selegiline less than 90 days prior to randomisation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BDI-IA total score | 12 weeks

SECONDARY OUTCOMES:
Evaluate if rasagiline compared to placebo improves cognitive function, over a treatment period of 12 weeks in idiopathic Parkinson´s Disease, using a formal neuropsychiatric cognitive test battery; quality of life (PDQ 39); apathy; ADL, motor function | 12 weeks
Change in quality of life using the PDQ-39 scale | 12 weeks
Change in apathy using the Apathy Scale | 12 weeks
Change in ADL and motor function using UPDRS scales part II and III, respectively | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (12):
- Italy (12):
  - IT010, Cagliari
  - IT007, Chieti
  - IT004, Genova
  - IT005, Lido di Camaiore
  - IT003, Messina
  - IT012, Milan
  - IT001, Naples
  - IT011, Roma
  - IT008, Rome
  - IT015, Torino
  - IT013, Venezia
  - IT009, Verona

REFERENCES:
- Available data/document: EMA EudraCT Results: 2009-011144-19 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2009-011144-19/results